CLINICAL TRIAL: NCT01559831
Title: Immune Responses to Revaccination After Potentially Insufficient Priming With the Japanese Encephalitis Vaccine IXIARO Batch JEV09L37
Brief Title: Immune Response in IXIARO Batch JEV09L37 Recipients Before and After Revaccination
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: IC51-319
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Japanese Encephalitis
Keywords: Japanese Encephalitis; IXIARO; Japanese Encephalitis Vaccine
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IXIARO (Other): IXIARO, applied according to licensed dose, intramuscular
  Interventions: Biological: IXIARO

INTERVENTIONS:
Biological: IXIARO — Vero-cell derived Japanese encephalitis (JE) vaccine IXIARO, 0.5 ml intramuscular

SUMMARY:
IC51-319 is a single-arm, open-label study that investigates immune responses in subjects undergoing revaccination after receiving the subpotent batch of IXIARO JEV09L37 during primary immunization.

DETAILED DESCRIPTION:
IC51-319 is a single-arm, open-label study that investigates immune responses in subjects undergoing revaccination after receiving the subpotent batch of IXIARO JEV09L37 during primary immunization.

A total of up to 50 subjects having received primary immunization of IXIARO batch JEV09L37 and who have not yet been revaccinated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years or older having received IXIARO batch JEV09L37 during primary immunization
* In female subjects, either childbearing potential terminated by surgery or 1 year post-menopausal, or a negative urine pregnancy test during screening and the willingness not to become pregnant during the entire study period by practicing reliable methods of contraception
* Written informed consent obtained from the subject prior to any study-related procedures

Exclusion Criteria:

* Vaccination against Yellow fever, Dengue Fever, West Nile Fever or TBE or vaccination with any JE vaccine since primary immunization with IXIARO JEC09L37
* Clinical manifestation of any flavivirus infection since primary immunization with IXIARO JEC09L37
* Acute febrile infections or exacerbation of chronic infection on the day of IXIARO vaccination
* Pregnancy, lactation or unreliable contraception in female subjects with child-bearing potential and unreliable contraception in male subjects.
* Use of any other investigational or non-registered drug within 30 days prior to the first vaccination with IXIARO Visit 1 and during the study period
* Any condition which might interfere with study objectives or would limit the subject's ability to complete the study in the opinion of the investigator
* Persons who are committed to an institution
* At Day 0, upcoming scheduled travel to a JE endemic region

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate (SCR) at Day 28 | at Day 28

SECONDARY OUTCOMES:
SCR at Day 0 | Day 0
Geometric Mean Titer at Day 0 and 28 | Day 0 and Day 28
Rate of Adverse Events up to Day 28 | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Vera Kadlecek, Mag., Study Chair — Valneva Austria GmbH
Locations (1):
- UCLH Foundation Trust, London, London, United Kingdom